CLINICAL TRIAL: NCT00492960
Title: A Phase IIb, Randomized, Double-Blind, Placebo Controlled, Dose Ranging, Multicenter Study to Determine the Safety, Tolerance, and Efficacy of Larazotide Acetate (AT-1001) in Celiac Disease Subjects During a Gluten Challenge
Brief Title: Study to Assess the Efficacy of Larazotide Acetate for the Treatment of Celiac Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 9 Meters Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLIN1001-006
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Celiac Disease
Keywords: larazotide acetate
MeSH Terms: conditions — Celiac Disease | interventions — larazotide acetate; Glutens

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo Controlled, dose ranging, multicenter Study
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Larazotide acetate 1 mg (Experimental): larazotide acetate 1 mg capsules TID + 900 mg gluten capsules TID for 6 weeks
  Interventions: Drug: larazotide acetate; Dietary Supplement: 900 mg gluten
- Larazotide acetate 4 mg (Experimental): larazotide acetate 4 mg capsules TID + 900 mg gluten capsules TID for 6 weeks
  Interventions: Drug: larazotide acetate; Dietary Supplement: 900 mg gluten
- Larazotide acetate 8 mg (Experimental): larazotide acetate 8 mg capsules TID + 900 mg gluten capsules TID for 6 weeks
  Interventions: Drug: larazotide acetate; Dietary Supplement: 900 mg gluten
- Placebo (Placebo Comparator): placebo capsules TID + 900 mg gluten capsules TID for 6 weeks
  Interventions: Drug: placebo; Dietary Supplement: 900 mg gluten

INTERVENTIONS:
Drug: larazotide acetate — gelatin capsules
  Other Names: AT-1001; INN-202
  Arms: Larazotide acetate 1 mg; Larazotide acetate 4 mg; Larazotide acetate 8 mg
Drug: placebo — gelatin capsules
  Arms: Placebo
Dietary Supplement: 900 mg gluten — gelatin capsules

SUMMARY:
This study was conducted to evaluate the efficacy of multiple doses of larazotide acetate in preventing intestinal permeability changes induced by a 6- week gluten challenge in subjects with celiac disease.

DETAILED DESCRIPTION:
This was a Phase IIb, randomized, double-blind, placebo-controlled, dose ranging, multicenter Study to determine the safety, tolerance, and efficacy of larazotide acetate in subjects with celiac disease during a gluten challenge. Subjects remained on their gluten-free diet throughout the duration of the trial. Study drug or drug placebo capsules were administered TID 15 minutes before each meal. Gluten or gluten placebo capsules will be taken TID with each meal.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults with biopsy proven celiac disease on a gluten-free diet for at least the past 6 months
* Anti-Tissue Transglutaminase (anti-tTG) ≤ 10 EU.
* BMI between 18.5 and 38, inclusive.

Exclusion Criteria

* Has chronic active GI disease other than celiac disease
* Has diabetes (Type 1 or Type 2).
* Unable to abstain from alcohol consumption or NSAID use for 48 hours prior to each intestinal permeability collection throughout the study.
* Has hemoglobin value below 8.5 g/dL

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2008-10 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of multiple doses larazotide acetate in preventing intestinal permeability changes induced by a 6- week gluten challenge. | Following ingestion of a solution of lactulose and mannitol; lactulose and mannitol excretion was quantified and the LAMA ratio calculated from overnight urine specimens collected on Days 7, 21, 35, 49 and 56.
  The primary efficacy endpoint was the Day 49 to Day 7 ratio of urinary LAMA ratios as a response to gluten

SECONDARY OUTCOMES:
Safety of a 6-week exposure to oral doses of larazotide acetate in celiac disease patients exposed to 900 mg gluten TID with meals | Up to 6 weeks
  Safety endpoints assessed in this study were adverse events, vital signs, physical examination results, clinical laboratory test results, concomitant medication usage and ECG results
To prospectively validate a composite, weighted index of celiac disease activity | GSRS was completed weekly throughout the study.
  Gastrointestinal symptoms were assessed by the GSRS patient self-assessment questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Leon, MD, Ph.D., Study Director — Alba Therapeutics Corp
Locations (23):
- United States (17):
  - Study Site, Scottsdale, Arizona
  - Study Site, Colorado Springs, Colorado
  - Study Site, Chicago, Illinois
  - Study Site, Lexington, Kentucky
  - Study Site, Hagerstown, Maryland
  - Study Site, Boston, Massachusetts
  - Study Site, Troy, Michigan
  - Study Site, Rochester, Minnesota
  - Study Site, New York, New York
  - Study Site, Asheville, North Carolina
  - Study Site, Cleveland, Ohio
  - Study Site, Philadelphia, Pennsylvania
  - Study Site, Pittsburgh, Pennsylvania
  - Study Site, Houston, Texas
  - Study Site, Plano, Texas
  - Study Site, Richmond, Virginia
  - Study Site, Seattle, Washington
- Canada (6):
  - Study Site, Edmonton, Alberta
  - Study Site, Kelowna, British Columbia
  - Study Site, Calgary
  - Study Site, Montreal
  - Study Site, Toronto
  - Study Site, Winnipeg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kelly CP, Green PH, Murray JA, Dimarino A, Colatrella A, Leffler DA, Alexander T, Arsenescu R, Leon F, Jiang JG, Arterburn LA, Paterson BM, Fedorak RN; Larazotide Acetate Celiac Disease Study Group. Larazotide acetate in patients with coeliac disease undergoing a gluten challenge: a randomised placebo-controlled study. Aliment Pharmacol Ther. 2013 Jan;37(2):252-62. doi: 10.1111/apt.12147. Epub 2012 Nov 19. PMID 23163616